CLINICAL TRIAL: NCT00005130
Title: Coronary Artery Risk Development in Young Adults (CARDIA)
Brief Title: Coronary Artery Risk Development in Young Adults
Acronym: CARDIA
Status: Active, not recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jing Li, Professor of Medicine, National Heart, Lung, and Blood Institute (NHLBI)
Other Study IDs: 1000
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Hypertension; Heart Diseases; Obesity; Diabetes Mellitus
Keywords: Cardiovascular Disease; Coronary Disease; Prospective Cohort Study; Longitudinal Observational Study
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Hypertension; Heart Diseases; Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, EDTA plasma, citrated plasma, urine, extracted DNA

SUMMARY:
To measure changes in coronary heart disease risk factors in cohorts of Black and White males and females 18 to 30 years of age at baseline. Also, to identify lifestyles during this age span which influence these changes in risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

Both epidemiologic and clinical research in coronary heart disease have increased our awareness that some risk factors for disease such as obesity, hypertension, and hypercholesterolemia may be partially determined by genetic factors or habits which are formed in infancy, childhood, and adolescence. Studies to date also suggest that some of the coronary heart disease risk factors do not change dramatically before the late teenage years and that differences in characteristics by sex or race are most pronounced after this time. However, relatively little work has been done to identify the characteristics of young adult life which may be precursors to or coincident with the increase in risk factors prior to middle age. While major increases in certain risk factors occur in young adulthood in conjunction with significant changes in life style, the interrelationships among these risk factors and changes have not been rigorously investigated.

Cross-sectional data, for example, suggest that weight gain is pronounced during the late teens through age 30, particularly in males, and that a linear relationship exists between weight and lipoprotein fractions at these ages. The reasons for and consequences of this increase in adiposity need further investigation. The interaction of life events, behavior, and changes in physical activity and dietary intake that may influence weight gain and lipoprotein concentrations should be determined, as well as the importance of weight gain in relationship to risk factor changes during this age span.

Investigators have examined the consistency of blood pressure levels in children to determine whether "tracking" occurs into the teenage years. The results of these studies have raised other interesting and important questions. Is there evidence for "tracking" of other coronary risk factors? Does "tracking" persist into young adult life, a time during which dramatic changes in life style are often taking place? The study will contribute to our understanding of the development of atherosclerosis and will help to determine an optimal strategy for prevention before individual life style patterns become well established. The Working Group on Heart Disease Epidemiology in 1978 recommended the study with highest priority. The study was approved by the National Heart, Lung, and Blood Advisory Council in November 1982. The Request for Proposals was released in December 1982.

DESIGN NARRATIVE:

CARDIA, which began recruitment in 1985, has completed 10 examinations in a cohort of 5,115 men and women aged 18-30 years in four communities in the US. Participants were initially sampled from the total population, selected census tracts or, in the case of one center, the membership of a large health plan. The original cohort had approximately equal representation by Black and White individuals, men and women, those aged 18-24 and 25-30 years, and those with no more than a high school education and more than a high school education. The baseline examination (Year 0) was conducted over a 14-month period during 1985-86. The examination consisted of questionnaires on sociodemographic characteristics, health behaviors, and psychological factors; an exercise treadmill test; resting electrocardiography; a diet history assessment; anthropometry; pulmonary function testing; and resting blood pressure. Fasting blood measurements included total cholesterol and its subfractions, insulin, glucose, liver enzymes and other serum chemistry measurements, and hematology.

Nine additional examinations have been completed every 2-5 years, including a Year 35 examination completed in 2022. Repeat measurements on traditional risk factors, including plasma lipids, blood pressure, anthropometry, smoking behavior, physical activity, and pulmonary function testing (except Years 7 and 15) have used the same methods at each examination to assess age and secular trends in these factors during young adulthood. In selected years, additional measurements have been made, including a treadmill exercise test at baseline, Year 7, Year 20, and Year 35 (in a subset); diet history at baseline, Year 7, Year 20, and Year 35 (in a subset); cardiovascular reactivity measurements in Year 2; echocardiography and ambulatory blood pressure monitoring at Year 5 (in a subset); skin reflectance and assessment of the experience of discrimination and other psychosocial measures and urine sodium and creatinine in Year 7; echocardiography (in a subset) in Year 10, glucose tolerance testing, and microalbuminuria in Year 10 and Year 20; coronary CT scan in Year 15 and Year 20; carotid intima media thickness in Year 20; and brain MRI (in a subset) in Years 25, 30, and 35.

Retention of the surviving cohort was 90, 86, 81, 79, 74, 72, 72, 71, and 71 percent at each of the respective follow-up examinations. Cohort members are contacted every six months to obtain information on vital status and current residence. Every other six-month contact also includes speaking with the participant to ascertain information on current smoking status, major illness or injury, and hospitalizations.

The Year 40 Exam will begin July 2026 and will continue through August 2027. There will be an estimated 2,994 participants from four field centers that will participate in this exam.

ELIGIBILITY:
Age 18-30 years, males and females, Black and White, free of long-term disease or disability that would interfere substantially with any part of the examination

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Black and White males and females 18 to 30 years of age at baseline (1985-1986).
Sampling Method: Non-Probability Sample
Enrollment: 5115 (Actual)
Dates: Start 1984-01; Primary Completion 2033-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease | baseline (1985) through 2033
  Incident coronary heart disease (fatal or nonfatal myocardial infarction, acute coronary syndrome without myocardial infarction, coronary revascularization, coronary heart disease death), stroke, heart failure, peripheral arterial disease

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T. Lackland, DrPH, Study Chair — Medical University of South Carolina; Jing Li, MD, DrPH, MS, Principal Investigator — University of Alabama at Birmingham; Cora E. Lewis, MD, MSPH, Principal Investigator — University of Alabama at Birmingham; Mercedes R Carnethon, PhD, Principal Investigator — Northwestern University; Ankeet S. Bhatt, MD, MBA, ScM, Principal Investigator — Kaiser Foundation Research Institute; Weihong J. Tang, MD, PhD, Principal Investigator — University of Minnesota

REFERENCES:
- [Background] For list of CARDIA publications, https://zenodo.org/communities/cardia-cc/records?q=&l=list&p=1&s=10&sort=newest
- [Derived] Hascher K, Brown R, Janulis P, Slone BR, Avila GV, Lewis CE, Schreiner PJ, Bhatt AS, Engle A, Beach LB, Rivera AS. Investigating Sex Differences in the Association of Disclosure and Concealment of Sexual Minority Identity With Cardiovascular Health in the CARDIA Cohort at Year 35. Biopsychosoc Sci Med. 2026 Jan 1;88(1):89-99. doi: 10.1097/PSY.0000000000001422. Epub 2025 Aug 12. PMID 40891748
- [Derived] Hao QY, Weng J, Zeng TT, Zeng YH, Guo JB, Li SC, Chen YR, Yang PZ, Gao JW, Li ZH. Dietary branched-chain amino acids intake and coronary artery calcium progression: insights from the coronary artery risk development in young adults (CARDIA) study. Eur J Nutr. 2025 Mar 19;64(3):131. doi: 10.1007/s00394-025-03649-2. PMID 40106011
- [Derived] Gao JW, Guo Q, Weng Y, Huang ZG, Zhang HF, Wu YB, Wang JF, Zhang SL, Liu PM. Predicting the risk of coronary artery calcium progression in the general population: insights from the MESA and CARDIA studies. Clin Radiol. 2025 Jan;80:106724. doi: 10.1016/j.crad.2024.10.006. Epub 2024 Oct 16. PMID 39546957
- [Derived] Gao JW, Hao QY, Lin Y, Li ZH, Huang ZG, Bai ZQ, Zhang HF, Wu YB, Xiong ZC, You S, Wang JF, Zhang SL, Liu PM. Variability in Lipid Profiles During Young Adulthood and the Risk of Coronary Artery Calcium Incidence in Midlife: Insights From the CARDIA Study. Circ Cardiovasc Imaging. 2024 Sep;17(9):e016842. doi: 10.1161/CIRCIMAGING.123.016842. Epub 2024 Sep 13. PMID 39268602
- [Derived] Xu X, Wang Z, Huang R, Guo Y, Xiong Z, Zhuang X, Liao X. Remnant Cholesterol in Young Adulthood Is Associated With Left Ventricular Remodeling and Dysfunction in Middle Age: The CARDIA Study. Circ Cardiovasc Imaging. 2023 Nov;16(11):e015589. doi: 10.1161/CIRCIMAGING.123.015589. Epub 2023 Nov 21. PMID 37988449
- [Derived] Nguyen HT, Vasconcellos HD, Keck K, Reis JP, Lewis CE, Sidney S, Lloyd-Jones DM, Schreiner PJ, Guallar E, Wu CO, Lima JAC, Ambale-Venkatesh B. Multivariate longitudinal data for survival analysis of cardiovascular event prediction in young adults: insights from a comparative explainable study. BMC Med Res Methodol. 2023 Jan 25;23(1):23. doi: 10.1186/s12874-023-01845-4. PMID 36698064
- [Derived] Hao QY, Gao JW, Yuan ZM, Gao M, Wang JF, Schiele F, Zhang SL, Liu PM. Remnant Cholesterol and the Risk of Coronary Artery Calcium Progression: Insights From the CARDIA and MESA Study. Circ Cardiovasc Imaging. 2022 Jul;15(7):e014116. doi: 10.1161/CIRCIMAGING.122.014116. Epub 2022 Jul 8. PMID 35861979
- [Derived] Heravi AS, Michos ED, Zhao D, Ambale-Venkatesh B, Doria De Vasconcellos H, Lloyd-Jones D, Schreiner PJ, Reis JP, Wu C, Lewis CE, Shikany JM, Sidney S, Guallar E, Ndumele CE, Ouyang P, Hoogeveen RC, Lima JAC, Vaidya D, Post WS. Oxidative Stress and Menopausal Status: The Coronary Artery Risk Development in Young Adults Cohort Study. J Womens Health (Larchmt). 2022 Jul;31(7):1057-1065. doi: 10.1089/jwh.2021.0248. Epub 2022 Jun 8. PMID 35675673
- [Derived] Gao JW, You S, Liu ZY, Hao QY, Wang JF, Vuitton DA, Zhang SL, Liu PM. Different Metabolic Phenotypes of Obesity and Risk of Coronary Artery Calcium Progression and Incident Cardiovascular Disease Events: The CARDIA Study. Arterioscler Thromb Vasc Biol. 2022 May;42(5):677-688. doi: 10.1161/ATVBAHA.122.317526. Epub 2022 Apr 7. PMID 35387482
- [Derived] Feng W, Zhang Z, Liu Y, Li Z, Guo W, Huang F, Zhang J, Chen A, Ou C, Zhang K, Chen M. Association of Chronic Respiratory Symptoms With Incident Cardiovascular Disease and All-Cause Mortality: Findings From the Coronary Artery Risk Development in Young Adults Study. Chest. 2022 Apr;161(4):1036-1045. doi: 10.1016/j.chest.2021.10.029. Epub 2021 Nov 2. PMID 34740593
- [Derived] Gao (高静伟) JW, Hao (郝卿鋆) QY, Zhang (张海峰) HF, Li (李雄志) XZ, Yuan (袁智敏) ZM, Guo (郭颖) Y, Wang (王景峰) JF, Zhang (张少玲) SL, Liu (刘品明) PM. Low-Carbohydrate Diet Score and Coronary Artery Calcium Progression: Results From the CARDIA Study. Arterioscler Thromb Vasc Biol. 2021 Jan;41(1):491-500. doi: 10.1161/ATVBAHA.120.314838. Epub 2020 Oct 29. PMID 33115269
- [Derived] Washko GR, Colangelo LA, Estepar RSJ, Ash SY, Bhatt SP, Okajima Y, Liu K, Jacobs DR Jr, Iribarren C, Thyagarajan B, Lewis CE, Kumar R, Han MK, Dransfield MT, Carnethon MR, Kalhan R. Adult Life-Course Trajectories of Lung Function and the Development of Emphysema: The CARDIA Lung Study. Am J Med. 2020 Feb;133(2):222-230.e11. doi: 10.1016/j.amjmed.2019.06.049. Epub 2019 Jul 29. PMID 31369720
- [Derived] Benck LR, Cuttica MJ, Colangelo LA, Sidney S, Dransfield MT, Mannino DM, Jacobs DR Jr, Lewis CE, Zhu N, Washko GR, Liu K, Carnethon MR, Kalhan R. Association between Cardiorespiratory Fitness and Lung Health from Young Adulthood to Middle Age. Am J Respir Crit Care Med. 2017 May 1;195(9):1236-1243. doi: 10.1164/rccm.201610-2089OC. PMID 28248551
- [Derived] Natarajan P, Young R, Stitziel NO, Padmanabhan S, Baber U, Mehran R, Sartori S, Fuster V, Reilly DF, Butterworth A, Rader DJ, Ford I, Sattar N, Kathiresan S. Polygenic Risk Score Identifies Subgroup With Higher Burden of Atherosclerosis and Greater Relative Benefit From Statin Therapy in the Primary Prevention Setting. Circulation. 2017 May 30;135(22):2091-2101. doi: 10.1161/CIRCULATIONAHA.116.024436. Epub 2017 Feb 21. PMID 28223407
- [Derived] Bantle AE, Chow LS, Steffen LM, Wang Q, Hughes J, Durant NH, Ingram KH, Reis JP, Schreiner PJ. Association of Mediterranean diet and cardiorespiratory fitness with the development of pre-diabetes and diabetes: the Coronary Artery Risk Development in Young Adults (CARDIA) study. BMJ Open Diabetes Res Care. 2016 Aug 31;4(1):e000229. doi: 10.1136/bmjdrc-2016-000229. eCollection 2016. PMID 27648287
- [Derived] Kirkegaard H, Nohr EA, Rasmussen KM, Stovring H, Sorensen TI, Lewis CE, Gunderson EP. Maternal prepregnancy waist circumference and BMI in relation to gestational weight gain and breastfeeding behavior: the CARDIA study. Am J Clin Nutr. 2015 Aug;102(2):393-401. doi: 10.3945/ajcn.114.099184. Epub 2015 Jul 1. PMID 26135344
- [Derived] Shikany JM, Jacobs DR Jr, Lewis CE, Steffen LM, Sternfeld B, Carnethon MR, Richman JS. Associations between food groups, dietary patterns, and cardiorespiratory fitness in the Coronary Artery Risk Development in Young Adults study. Am J Clin Nutr. 2013 Dec;98(6):1402-9. doi: 10.3945/ajcn.113.058826. Epub 2013 Oct 2. PMID 24088719
- [Derived] Ogunyankin KO, Liu K, Lloyd-Jones DM, Colangelo LA, Gardin JM. Reference values of right ventricular end-diastolic area defined by ethnicity and gender in a young adult population: the CARDIA study. Echocardiography. 2011 Feb;28(2):142-9. doi: 10.1111/j.1540-8175.2010.01290.x. Epub 2011 Jan 7. PMID 21210835
- [Derived] Kalhan R, Tran BT, Colangelo LA, Rosenberg SR, Liu K, Thyagarajan B, Jacobs DR Jr, Smith LJ. Systemic inflammation in young adults is associated with abnormal lung function in middle age. PLoS One. 2010 Jul 2;5(7):e11431. doi: 10.1371/journal.pone.0011431. PMID 20625390
- [Derived] Bibbins-Domingo K, Pletcher MJ, Lin F, Vittinghoff E, Gardin JM, Arynchyn A, Lewis CE, Williams OD, Hulley SB. Racial differences in incident heart failure among young adults. N Engl J Med. 2009 Mar 19;360(12):1179-90. doi: 10.1056/NEJMoa0807265. PMID 19297571
- See also: CARDIA public website — https://sites.uab.edu/cardia/
- Available data/document: Individual Participant Data Set: CARDIA — http://biolincc.nhlbi.nih.gov/studies/cardia/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — https://sites.uab.edu/cardia/for-researchers/exam-materials/protocols/
- Available data/document: Informed Consent Form — https://sites.uab.edu/cardia/for-researchers/exam-materials/consent-forms/
- Available data/document: Data Collection Forms — https://sites.uab.edu/cardia/for-researchers/exam-materials/data-collection-forms/
- Available data/document: Study Manuals — https://sites.uab.edu/cardia/for-researchers/exam-materials/manuals-of-operation/